CLINICAL TRIAL: NCT06625541
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Ascending Doses of AJ302-IM in Healthy Volunteers Via Intramuscular Injection
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AJ302-IM in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AnnJi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: AJ79009-302IM-101
Record Dates: First submitted 2024-08-14; First posted 2024-10-03 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AJ302-IM (Experimental)
  Interventions: Drug: AJ302-IM
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AJ302-IM — 7 cohorts (7 dose levels) of participants are planned to be dosed.
  Arms: AJ302-IM
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of AJ302-IM following intramuscular administration of single ascending doses in healthy volunteers.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female, non-smokers (no use of tobacco or nicotine products within 3 months prior to screening), ≥ 18 and ≤ 55years of age, with body mass index (BMI) ≥ 18.5 and ≤ 30.0 kg/m2 and body weight ≥ 50.0 kg for males and ≥ 45.0 kg for females.
* Normal renal function at screening.
* Healthy as defined by:

  * The absence of clinically significant illness and surgery within 4 weeks prior to study drug administration.
  * The absence of clinically significant history of neurological, endocrine, cardiovascular, respiratory, hematological, immunological, psychiatric, depression, attempted suicide, gastrointestinal, renal, hepatic, and metabolic disease.
* Able to understand the study procedures and provide signed informed consent to participate in the study

Key Exclusion Criteria:

* Any clinically significant abnormal finding at physical examination
* Any lifetime suicidal behavior or suicidal ideation of type 4 (active suicidal ideation with some intent to act, without specific plan) or type 5 (active suicidal ideation with specific plan and intent) in the 2 years before screening based on the C-SSRS
* Clinically significant abnormal laboratory test results or positive serology test results for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV) antigen and antibody, at screening
* Positive pregnancy test or lactating female volunteers
* Positive urine drug screen, urine cotinine test, or alcohol breath test at screening and on Day -1
* History of significant allergic reactions to any drug
* Known allergy or hypersensitivity to histone deacetylase 6 (HDAC6) inhibitors or its derivatives and/or any study product excipients
* Clinically significant ECG abnormalities or vital signs abnormalities at screening
* History of drug abuse or recreational use of soft drugs or hard drugs
* History of alcohol abuse
* History of smoking or uses other nicotine-containing products
* Undergone major surgery ≤ 2 months before study drug administration
* History of clinically significant opportunistic infection or serious local infection or significant medical/surgical procedure or trauma, or any current infection.
* Use of medications for the timeframes specified in the protocol
* Received any investigational drug or any investigational device or any biological product within the timeframes specified in the protocol
* Tattoos, sunburn, scarring or anything that may interfere with evaluation of the injection site

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2024-06-24 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Incidence and proportion of volunteers with AEs including TEAEs and SAEs | Baseline up to Day 57

SECONDARY OUTCOMES:
Plasma PK of AJ302-IM | Pre-dose to Day 57
  AUC0-168hr: Area under the plasma concentration-time curve from zero to 168 hours
Plasma PK of AJ302-IM | Pre-dose to Day 57
  AUC0-inf: Area under the concentration-time curve from time zero to infinity (extrapolated)
Plasma PK of AJ302-IM | Pre-dose to Day 57
  AUC0-last: Area under the plasma concentration-time curve from zero to the last observed concentrations
Plasma PK of AJ302-IM | Pre-dose to Day 57
  Cmax: Maximal observed concentration
Plasma PK of AJ302-IM | Pre-dose to Day 57
  Tmax: Time when the maximal concentration is observed
Plasma PK of AJ302-IM | Pre-dose to Day 57
  Residual area: Percentage of AUC0-inf due to extrapolation from the time of the last observed concentration to infinity, calculated as [1 (AUC0 last/AUC0-inf)] x 100
Plasma PK of AJ302-IM | Pre-dose to Day 57
  T½ el: Terminal elimination half-life
Plasma PK of AJ302-IM | Pre-dose to Day 57
  Kel: Terminal elimination rate constant
Plasma PK of AJ302-IM | Pre-dose to Day 57
  Cl/F: Apparent clearance
Plasma PK of AJ302-IM | Pre-dose to Day 57
  Vz/F: Apparent volume of distribution
Urine PK of AJ302-IM | Pre-dose to Day 8
  Ae0-168hr: Cumulative urinary excretion from time zero to 168 hours, calculated as the sum of the amounts excreted over each collection interval
Urine PK of AJ302-IM | Pre-dose to Day 8
  Rmax: Maximal rate of urinary excretion, calculated by dividing the amount of drug excreted in each collection interval by the time over which it was collected
Urine PK of AJ302-IM | Pre-dose to Day 8
  TRmax: Time of maximal urinary excretion, calculated as the midpoint of the collection interval during which Rmax occurred
Urine PK of AJ302-IM | Pre-dose to Day 8
  ClR: Renal clearance, calculated as Ae0-168hr /AUC0-168hr

CONTACTS AND LOCATIONS:
Locations (1):
- AnnJi Investigational Site, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No